CLINICAL TRIAL: NCT01396356
Title: Impact of Atrial Fibrillation Ablation on Gastric Motility "The AF Gut Study"
Brief Title: Atrial Fibrillation Ablation on Gastric Motility "The AF Gut Study"
Status: Completed | Type: Observational
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Associate Professor of Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 12164
Record Dates: First submitted 2011-06-20; First posted 2011-07-18 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Atrial Fibrillation Ablation Procedure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ablation procedure
  Interventions: Procedure: GI procedures

INTERVENTIONS:
Procedure: GI procedures — If you agree to participate in the study, you will undergo a series of tests about a week before the expected ablation procedure. The same tests will be repeated 24-48 hours after the ablation. These tests include esophageal manometry, gastric emptying scan, sham feeding test and completing a symptoms questionnaire.

SUMMARY:
You are being scheduled to undergo an ablation procedure to treat your atrial fibrillation. Complications of ablation procedures include damage to structures near the heart from the heat energy used during the ablation procedure. These complications include damage to the esophagus (the tube through which food passes when you swallow) and stomach. A rare but often fatal complication resulting from severe heat damage is called an atrio-esophageal fistula (an abnormal connection between the heart and esophagus). However, the frequency of minimal damage to the esophagus or nerves of the gut that may go unnoticed are not known.

This study is designed to determine how often atrial fibrillation ablation causes problems with the stomach and esophagus.

ELIGIBILITY:
Inclusion criteria:

* All patients aged 18 years or more who undergo pulmonary vein isolation with radiofrequency ablation for clinically indicated atrial fibrillation.

Exclusion criteria:

1. Patients with established diagnosis of esophageal or gastric function abnormalities.
2. Patients who are unable to give consent or major psychiatric condition not under control.
3. Patients who had abdominal surgical procedures on stomach, esophagus or pancreas (Esophagectomy, Gastrostomy, Gastrectomy (Billroth I, Billroth II, Roux-en-Y), Bariatric surgery [Gastric bypass surgery, Adjustable gastric band, Sleeve gastrectomy, Vertical banded gastroplasty surgery], Gastroenterostomy, Hill repair, Nissen fundoplication, Gastropexy, Pancreatectomy, Pancreaticoduodenectomy, Pancreas transplantation, vagotomy).
4. Patients who unable to undergo any of the above mentioned procedures namely, esophageal manometry or sham feeding test or scientigraphy gastric emptying scan.
5. Patients with chronic pancreatitis.
6. Patients with either acute or chronic neuropathies such as diabetic, inflammatory, autoimmune and cranial neuropathies effecting vagal nerve or gastroparesis or achalasia. Limited peripheral neuropathies such as carpal tunnel syndrome or isolated Bell's palsy can be included.
7. Patients who have undergone previous radiofrequency ablation for atrial fibrillation or patients who had history of either minimally invasive or invasive or maze or modified maze procedures for atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: If you agree to participate in the study, you will undergo a series of tests about a week before the expected ablation procedure. The same tests will be repeated 24-48 hours after the ablation. These tests include esophageal manometry, gastric emptying scan, sham feeding test and completing a symptoms questionnaire.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine if pulmonary vein isolation with radiofrequency ablation impacts the upper gastrointestinal function by evaluating the Gastric and esophageal motility the lower esophageal sphincter tone changes by esophageal manometry. | up to 2 weeks
  The esophageal body motility is measured by recording the response to at least 10 wet swallows of 5-10 ml volume.

SECONDARY OUTCOMES:
To determine if pulmonary vein isolation with radiofrequency ablation impacts the upper gastrointestinal function by evaluating the Gastric and esophageal motility gastric emptying time measured by a scintigraphy gastric emptying scan. | up to 2 weeks
  Anterior and posterior scintigraphic images of the stomach will be obtained within 1 minute of completion of the meal (defined as 0) and at 60, 120, 180, and 240 minutes.
To determine if pulmonary vein isolation with radiofrequency ablation impacts the upper gastrointestinal function by evaluating the Gastric and esophageal motility through the vagal nerve function by sham feeding test. | up to 2 weeks
  Blood samples of glucose and pancreatic polypeptide will be collected at 10-minute intervals for 30 minutes after the initiation of the meal. If the elevation over baseline value of pancreatic polypeptide after the sham meal is <50%, then this is considered as a positive test, indicating that vagal nerve damage or essentially that a "vagotomy" had occurred.
To determine if pulmonary vein isolation with radiofrequency ablation impacts the upper gastrointestinal symptoms measured by serial upper GI questionnaire (PAGI-SYM®) scores. | up to 3 months
  The questionnaire has good reproducibility for measuring GI symptoms and validated. The questionnaire will be used at baseline at 3 months after PVI ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Lakkireddy D, Reddy YM, Atkins D, Rajasingh J, Kanmanthareddy A, Olyaee M, Dusing R, Pimentel R, Bommana S, Dawn B. Effect of atrial fibrillation ablation on gastric motility: the atrial fibrillation gut study. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):531-6. doi: 10.1161/CIRCEP.114.002508. Epub 2015 Mar 14. PMID 25772541